CLINICAL TRIAL: NCT00348504
Title: Survival of Patients With Acute Heart Failure in Need of Intravenous Inotropic Support: a Multicentre, Parallel-Group, Randomised, Double-Blind, Double-Dummy Study of Levosimendan Versus Dobutamine in Patients With Acute Heart Failure.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3001077
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Simendan; Dobutamine

INTERVENTIONS:
Drug: levosimendan
Drug: dobutamine

SUMMARY:
The primary objective of the study is to compare the efficacy of levosimendan and dobutamine on all-cause mortality in the 180 days following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed and dated informed consent
* Male and female patients over 18 years of age. Females of childbearing potential must have a negative pregnancy test and must refrain from breastfeeding. Women who are postmenopausal [two years since last menstrual cycle], surgically sterilised or who have undergone a hysterectomy are considered not to be of childbearing potential
* Hospitalised patients with acutely decompensated heart failure
* Left ventricular ejection fraction less than or equal to 30 % as assessed using echocardiography, radionuclide ventriculography or contrast angiography within 12 months
* Clinical need for intravenous inotropic support as evidenced by insufficient response to intravenous diuretics and/or vasodilators (nitroglycerin, nitroprusside) and at least one of the following at screening:

  * oliguria (mean urine output < 30 ml/h for at least 6 hours) and not a result of hypovolemia
  * dyspnoea at rest or mechanical ventilation for heart failure
  * haemodynamic impairment in those patients with Swan-Ganz catheter inserted (PCWP ≥ 18 mmHg and/or Cardiac Index ≤ 2.2 l/min/m2)

Exclusion Criteria:

* Severe obstruction of ventricular outflow tracts such as haemodynamically significant uncorrected primary valve disease or hypertrophic cardiomyopathy or impaired ventricular filling such as restrictive cardiomyopathy
* Weight ≥ 160 kg
* Cardiac surgery within 30 days before screening
* Stroke within 3 months before screening
* Systolic blood pressure persistently less than 85 mmHg at screening or at baseline
* Heart rate persistently 130 bpm or greater at screening or at baseline
* Serum potassium less than 3.5 mmol/l at screening
* Administration of any inotropic agent (e.g. dobutamine, milrinone, amrinone, enoximone, epinephrine, norepinephrine) except digitalis or dopamine (with dose of less than or equal than 2 mg/kg/min) during the current hospitalisation
* Hypersensitivity to levosimendan or dobutamine or any of their excipients
* A history of Torsades de Pointes
* Severe renal insufficiency (serum creatinine > 450 mmol/l [5.0 mg/dl]) or on dialysis
* Significant hepatic impairment at discretion of the investigator
* Acute bleeding
* Severe anemia (haemoglobin < 8 g/dl) at screening
* Septicaemia or septic shock
* Other serious diseases limiting life expectancy considerably (e.g. end-stage cancer)
* Participation in a clinical trial with any experimental treatment within 30 days prior to screening or previous participation in the present study
* Administration of levosimendan within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300
Dates: Start 2003-03; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
All-cause mortality in the 180 days following randomization.

SECONDARY OUTCOMES:
All-cause mortality during the 31 days following randomization
Mean change in plasma BNP concentration from baseline to 24 hours after the start of the study drug infusion
Number of day alive and out of hospital (DAOH) during the 180 days following randomization
Patient's evaluation of change in dyspnea at 24 hours following randomization
Patient's evaluation of change in Global Assessment at 24 hours following randomization
Cardiovascular mortality during the 180 days following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Padley, M.D., Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, Abbott Park, Illinois, United States

REFERENCES:
- [Derived] Cohen-Solal A, Logeart D, Huang B, Cai D, Nieminen MS, Mebazaa A. Lowered B-type natriuretic peptide in response to levosimendan or dobutamine treatment is associated with improved survival in patients with severe acutely decompensated heart failure. J Am Coll Cardiol. 2009 Jun 23;53(25):2343-8. doi: 10.1016/j.jacc.2009.02.058. PMID 19539144
- [Derived] Mebazaa A, Nieminen MS, Packer M, Cohen-Solal A, Kleber FX, Pocock SJ, Thakkar R, Padley RJ, Poder P, Kivikko M; SURVIVE Investigators. Levosimendan vs dobutamine for patients with acute decompensated heart failure: the SURVIVE Randomized Trial. JAMA. 2007 May 2;297(17):1883-91. doi: 10.1001/jama.297.17.1883. PMID 17473298